CLINICAL TRIAL: NCT05168566
Title: A Multicenter, Open-label, Phase IIb Study to Evaluate the Efficacy and Safety of Sutetinib Maleate Capsule in Locally Advanced or Metastatic NSCLC (Non-resistant Uncommon EGFR Mutations Only, Including L861Q, G719X, and/or S768I)
Brief Title: Study to Evaluate Sutetinib Maleate Capsule in Locally Advanced or Metastatic Non-small Cell Lung Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Teligene US (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SZCT-2020-06
Record Dates: First submitted 2021-12-12; First posted 2021-12-23 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Malignant tumor; EGFR mutation; lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasms; Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Sutetinib Maleate Arm (Experimental): Sutetinib capsules monotherapy
  Interventions: Drug: Sutetinib Maleate Capsule

INTERVENTIONS:
Drug: Sutetinib Maleate Capsule — Study drug to be taken orally with or without food (with food preferred) for up to13 cycles
  Other Names: Sutetinib

SUMMARY:
This is a Phase 2b, multicenter, open-label study to evaluate the safety and efficacy of Sutetinib Maleate Capsule in Locally Advanced or Metastatic NSCLC (Non-resistant Uncommon EGFR Mutations Only, Including L861Q, G719X, and/or S768I)

DETAILED DESCRIPTION:
Sutetinib is an investigational irreversible EGFR tyrosine kinase inhibitor. EGFR is a gene that makes a protein that is involved in cell growth and cell survival. Mutated (changed) forms of the EGFR gene and protein have been found in some types of cancer, including non-small cell lung cancer. These changes may cause cancer cells to grow and spread in the body. The purpose of this study is to explore how effective Sutetinib maleate capsules are for the treatment of patients with locally advanced or metastatic NSCLC with non-resistant uncommon EGFR mutations

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years old and above, male or female.
2. Histopathological and/or cytopathological confirmation of locally advanced or metastatic NSCLC patients with ≤ 1 prior line of chemotherapy.
3. Confirmation that the tumor harbors a non-resistant uncommon EGFR mutation (tumor tissue biopsy), including one or more of L861Q, G719X and S768I mutations, excluding any other EGFR sensitive mutations and/or oncogenes..
4. At least one measurable lesion.
5. ECOG score of 0, 1, or 2.
6. A minimum life expectancy of > 3 months.
7. Adequate bone marrow reserve, hepatic, renal and coagulation function.
8. Willingness of all subjects of childbearing potential to use acceptable methods of birth control.

Exclusion Criteria:

1. Ever used the epidermal growth factor receptor-tyrosine kinase inhibitor (EGFR-TKI) for anti-tumor therapy prior to enrollment.
2. Any systemic anti-tumor therapy such as chemotherapy, immunotherapy and radiation therapy used within 4 weeks prior to enrollment; any palliative radiotherapy for non-target lesions used to relieve symptoms and traditional Chinese medicines indicated for tumor within 2 weeks prior to enrollment.
3. Use or intake of drugs or foods containing potent inhibitor or inducer of cytochrome P450 isozyme 3A4 (CYP3A4) within 14 days or 5 half-lives, whichever was the longer, prior to enrollment.
4. Surgical operation (excluding aspiration biopsy) of main organs or a significant injury within 4 weeks prior to enrollment.
5. Any unresolved toxicities from prior therapy greater than Grade 1 at the time of screening except alopecia.
6. Inability to swallow the study medication, any seriously chronic gastrointestinal disorder, malabsorption syndrome or any other conditions with influence on gastrointestinal absorption.
7. Active central nervous system metastases
8. Previous or current interstitial lung disease, radiation pneumonitis which requires hormone therapy, or drug-related pneumonia, idiopathic interstitial pulmonary fibrosis identified in a baseline CT scan; uncontrolled massive pleural or pericardial effusion.
9. Any active infection which has not been controlled at screening.
10. Any serious cardiovascular disease.
11. History of other serious systemic disease not suitable for clinical trial.
12. Participation in other interventional clinical trial 4 weeks prior to enrollment or within 5 half-lives from the last dose of investigational product (whichever is longer).
13. Known alcohol or drug dependence.
14. Mental disorders or poor compliance.
15. Previously received solid organ transplantation or hematopoietic stem cell transplantation.
16. Females who are pregnant or breastfeeding.
17. Known hypersensitivity to the active ingredients or excipients of the investigational product.
18. Have any other primary malignant tumors within 3 years (except some low- risk cancers).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Assessment of Objective response rate (ORR) | 2 Years
  Objective response rate (ORR) assessed by IRC

SECONDARY OUTCOMES:
Assessment of Duration of response (DoR) | 2 Years
Assessment of Disease control rate (DCR) | 2 Years
Assessment of Progression free survival (PFS) | 2 Years
Assessment of Time to progressive disease | 2 Years
Assessment of Time to response | 2 Years
Assessment of Time to treatment failure (TTF) | 2 Years
Assessment of Overall survival (OS) | 2 Years
Assessment of 1-year progression-free survival | 1 Year
Assessment of 1-year survival | 1 Years
Assess incidence of Treatment-Emergent Adverse Events [Safety and Tolerability]). | 2 Years
  Safety and tolerability as determined by the incidence of adverse events (AEs), including severe AEs and serious AEs(SAEs)
Assessment of Peak Plasma Concentration (Cmax) or Area under the plasma concentration versus time curve (AUC) | 2 Years

CONTACTS AND LOCATIONS:
Locations (26):
- United States (6):
  - OPN Healthcare, Inc., Glendale, California
  - University Cancer & Blood Center, Athens, Georgia
  - Baptist Health, Louisville, Kentucky
  - University of Maryland Medical Center, Baltimore, Maryland
  - FirstHealth Cancer Center, Pinehurst, North Carolina
  - The University of Texas- MD Anderson Cancer Center, Houston, Texas
- China (20):
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Beijing Chest Hospital, Beijing, Beijing Municipality
  - The Affiliated Cancer Hospital of Chongqin University, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Wuhan Union Hospital of China, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Jilin Cancer Hospital, Changchun, Jilin
  - The First Affiliated Hospital of China Medical University, Shengyang, Liaoning
  - Linyi Cancer Hospital, Linyi, Shangdong
  - Shanghai Chest Hospital, Shanghai, Shanghai Municipality
  - Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality
  - Sichuan Cancer Hospital, Chengdu, Sichuan
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No